CLINICAL TRIAL: NCT01315080
Title: Efficacy of Percutaneous Injection of Triamcinolone in the Treatment of Mammillary Fistula
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitario Virgen de la Arrixaca (Other)
Responsible Party: Juan de Dios Berna Serna, MD PhD, Virgen de la Arrixaca University Hospital
Other Study IDs: FISTULA001
Record Dates: First submitted 2011-03-11; First posted 2011-03-15 (Estimated); Last update posted 2011-03-15 (Estimated); Status verified 2011-03

CONDITIONS: Mammillary Fistula
Keywords: mammillary fistula; triamcinolone; ultrasound management; percutaneous treatment

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Saline: Percutaneous drainage and saline solution irrigation
- Triamcinolone: Percutaneous drainage and saline solution irrigation plus percutaneous triamcinolone

SUMMARY:
The investigators recently proposed a new hypothesis on the pathogenesis of mammillary fistulae (MF) suggesting that occlusion of hair follicles by keratinous plugging may relevantly contribute to the development of MF. The investigators believe that the pathogenesis of MF mimics the behaviour of hidradenitis suppurative, as both clinical entities manifest themselves as a chronic, suppurative and recurrent inflammatory process. This new proposal has led to the present suggestion of a therapeutic alternative for MF.

DETAILED DESCRIPTION:
To compare the results from a prospective observational database with two groups of patients:

1. patients with MF treated by percutaneous drainage and saline solution.
2. patients with MF treated by percutaneous drainage and saline solution plus percutaneous triamcinolone.

These patients are treated following usual clinical practice in our Department. All the procedures are made through an ultrasound-guided way. During the follow-up of these cases (clinical and with ultrasound) resolution rate will be registered by the same investigator.

The follow-up will be at least 6 months.

ELIGIBILITY:
Inclusion Criteria:

* mammillary fistula
* older than 18 years
* patient acceptation to the recruitment

Exclusion Criteria:

* diabetes mellitus
* arterial hypertension
* immunodepression
* peptic ulcer
* chronic bowel inflammatory diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mammillary fistula
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-03 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Resolution of mammillary fistula | one year

CONTACTS AND LOCATIONS:
Overall Officials: Juan D Berna, MD PhD, Principal Investigator — Virgen de la Arrixaca University Hospital
Locations (1):
- Virgen de la Arrixaca University Hospital, Murcia, Murcia, Spain